CLINICAL TRIAL: NCT04082988
Title: Early Response Evaluation With 18F-FDG PET/CT and Immunological Profiling of Circulating Immune Cells and Tumor-draining Lymph Nodes in Non-small Cell Lung Cancer Patients Treated With Immunotherapy.
Brief Title: Early Response Evaluation in NSCLC Patients Treated With Immunotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been closed due to slow enrollment.
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M17IPL
Record Dates: First submitted 2018-11-09; First posted 2019-09-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: NSCLC, Stage IV
Keywords: PD-L1 expression; eligible for treatment with nivolumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Other): Nivolumab treatment according to label: 3 mg/kg nivolumab IV Q2W, 240mg Q2W or 480mg Q4W as an IV infusion until disease progression or unacceptable toxicity.
  FDG PET-CT will be performed at baseline and between 7 and 14 days after treatment initiation
  Interventions: Diagnostic Test: 18F-FDG PET-CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET-CT — 18F-FDG PET-CT scan
  Other Names: Tracer

SUMMARY:
A pilot study with biomarker exploration.50 patients with stage IV non-small cell lung cancer (NSCLC) that are eligible for treatment with nivolumab. Patients will undergo a 18F-FDG-PET/CT and EBUS-FNA of the lymph nodes and have blood drawn before and after immune checkpoint inhibitor treatment to compare tumor FDG uptake and to identify changes in the immune effector cell subsets in TDLNs. Blood will be drawn in parallel to compare the distribution of immune effector cell subsets before and after treatment initiation. Because of the possible burden for patients, the EBUS-FNA is not mandatory to complete the study and is there for an exploratory objective. Also blood will be drawn for a tumor mutational burden at baseline. The first six patients will undergo a dynamic PET-CT scan in addition to a static scan to study the influence of possible immunotherapy induced changes to the body distribution and kinetics of FDG..

DETAILED DESCRIPTION:
Early response evaluation with 18F-FDG PET/CT and immunological profiling of circulating immune cells and tumor-draining lymph nodes in non-small cell lung cancer patients treated with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide written informed consent for the study.
* ≥ 18 years of age on day of signing informed consent.
* confirmed diagnosis of NSCLC.
* Histological tumor biopsy for PD-L1 IHC assessment (DAKO assay) available.
* Ipsilateral hilar or mediastinal lymph node with a short axis diameter ≥1 cm.
* Eligible and planned to receive nivolumab according to EMA label and national guidelines.
* Measurable disease according to RECIST v1.1.
* WHO performance status of 0-2.

Exclusion Criteria:

* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to baseline PET-scan.
* Has an active infection or had an active infection within 2 weeks prior to baseline PET-scan.
* Has a known history of hypersensitivity to contrast material.
* Isolated distant relapse after curative intent treatment for stage I-III NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Percentage of collected immune cells by FNA EBUS will be assesed using flow cytometry. | Baseline and at the end of cycle 1 (each cycle is 14 days).
  The change in the percentages of selected immune cell parameters (CD4+ T, CD8+ T cells) after immunotherapy treatment as compared to baseline will be calculated
Percentage of collected immune cells by FNA EBUS will be assesed using flow cytometry. | Baseline and at the end of cycle 1 (each cycle is 14 days).
  The change in the percentages of selected immune cell parameters (CD8+ T cells) after immunotherapy treatment as compared to baseline will be calculated
FDG PET-CT analysis | Baseline and at the end of cycle 1 (each cycle is 14 days).
  Parameter change (SUVpeak) between both scans will be measured.
FDG PET-CT analysis | Baseline and at the end of cycle 1 (each cycle is 14 days).
  Parameter change (SUVmax) between both scans will be measured.
FDG PET-CT analysis | Baseline and at the end of cycle 1 (each cycle is 14 days).
  Parameter change (SUVmean) between both scans will be measured.
Peripheral blood mononuclear cells will be isolated and counted using FACS | Baseline and at the end of cycle 1 (each cycle is 14 days).
  PBMC's will be counted at two timepoints. Change between both timepoints will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: J de Langen, MD, PhD, Principal Investigator — NKI-AvL
Locations (2):
- Netherlands (2):
  - VU medical center, Amsterdam
  - Leiden University Medical Center, Leiden

IPD SHARING:
Plan to Share IPD: Undecided
to be decided

REFERENCES:
- [Derived] Borm FJ, Smit J, Bakker J, Wondergem M, Smit EF, de Langen AJ, de Gruijl TD. Early response evaluation of PD-1 blockade in NSCLC patients through FDG-PET-CT and T cell profiling of tumor-draining lymph nodes. Oncoimmunology. 2023 Apr 26;12(1):2204745. doi: 10.1080/2162402X.2023.2204745. eCollection 2023. PMID 37123045